CLINICAL TRIAL: NCT04618497
Title: A Pilot Study on the Use of Methoxyflurane (Penthrox®) for Pain Control in the Emergency Department
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Wong Ka Ying, Medical Officer, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKECREC-2020-064
Record Dates: First submitted 2020-10-23; First posted 2020-11-06 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Traumatic Pain
MeSH Terms: interventions — Methoxyflurane; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled on a convenience basis. After being seen and screened by investigators, patients who meet all inclusion and non-exclusion criteria will be enrolled and randomized 1:1 by drawing from equal preset numbers of envelopes. Patients will receive either inhalational methoxyflurane or intramuscular ketorolac. Patients and investigators are not blinded to the treatment due to the nature of drug administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalational methoxyflurane (Penthrox) (Experimental)
  Interventions: Drug: Methoxyflurane
- Intramuscular ketorolac (Active Comparator)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Methoxyflurane — Each patient in the methoxyflurane group will use one Penthrox inhaler under supervision of trained personnel. After priming the inhaler with 3 mL of methoxyflurane, patient is instructed to inhale through the mouthpiece to obtain analgesia, and then exhale back into the mouthpiece so that any unmetabolized methoxyflurane can be adsorbed by activated charcoal chamber. First few breaths should be gentle and then breathe normally through Inhaler. Onset of pain relief is rapid and occurs after 6-10 inhalations. If stronger analgesia is required, patient can cover the diluter hole with a finger during inhalation. Patients are able to titrate the amount of methoxyflurane inhaled and should be instructed to inhale intermittently to achieve adequate pain control.
  Other Names: Penthrox
  Arms: Inhalational methoxyflurane (Penthrox)
Drug: Ketorolac — Each patient in the ketorolac group will receive one dose of 30mg intramuscular ketorolac injected at gluteal muscle by nursing staff as usual daily practice.
  Other Names: Toradol
  Arms: Intramuscular ketorolac

SUMMARY:
Patients commonly visit the emergency department (ED) for pain after musculoskeletal injury and need early treatment with analgesic. Prompt and adequate pain relief can reduce suffering and promote early discharge and return to work. Nonsteroidal anti-inflammatory drugs (NSAIDs) and opioids are the major injectable analgesic used for moderate to severe pain in EDs in Hong Kong. They are given via intravenous or intramuscular route for faster onset of action to achieve rapid pain relief in the emergency setting. However, injections are invasive and can be distressing for patients. Methoxyflurane (Penthrox®) is recently introduced to our emergency department as an inhalational analgesic. It has been granted registration approval in Hong Kong since 2018, but it is not widely used in the locality. Methoxyflurane is a volatile fluorinated hydrocarbon self-administrated by inhalation through a portable hand-held whistle-shaped inhaler device (Penthrox®) to relieve pain associated with trauma or minor surgical procedures in stable and conscious patients. In this study, the investigators will evaluate the efficacy and safety Penthrox® in the treatment of acute traumatic pain in hospital emergency department setting by comparing it to another conventional analgesic commonly used.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes from 18 to 64 years of age
* Presented to the ED in Ruttonjee Hospital for musculoskeletal injury within 72 hours of onset (Types of injury include contusion, sprain, crushing, burn, laceration, fracture and dislocation)
* Moderate pain at screening (10-point Numeric Rating Scale ≥4 to ≤7)

Exclusion Criteria:

* Critical or life-threatening condition requiring resuscitation
* Limb-threatening condition or any injuries requiring immediate management
* Hemodynamically unstable (systolic blood pressure <90 mmHg, diastolic blood pressure <60mmHg)
* Respiratory distress with respiratory rate >20 breath per minute or oxygen saturation <95% on room air
* Pregnant or breastfeeding women
* Impaired consciousness from any cause such as head injury and acute intoxication, based on the judgement of investigator
* Any physical, visual or cognitive conditions that may affect patient's ability to use visual analog scale for self-assessments of pain intensity
* Concomitant use of other analgesic within 5 hours (8 hours for diclofenac sodium) prior to presentation to ED
* Other pre-existing chronic pain condition
* Unable or refuse to provide written informed consent
* Unable to understand and converse in the language spoken
* Contraindication to inhalational methoxyflurane

  1. Known personal or family history of hypersensitivity to methoxyflurane or any fluorinated anesthetics
  2. Known pre-existing clinically significant renal or hepatic impairment
  3. Known personal or family history of malignant hyperthermia
  4. Concomitant use of nephrotoxic agents such as gentamicin, tetracycline, colistin, polymyxin B and amphotericin B
  5. Concomitant use of cytochrome P450 inducers such as alcohol, isoniazid, phenobarbital and rifampicin
* Contraindication to intramuscular ketorolac

  1. Known allergy to NSAIDS
  2. Known pre-existing clinically significant renal impairment or at risk for renal failure due to volume depletion
  3. Active major bleeding
  4. Suspected or confirmed cerebrovascular bleeding
  5. History of peptic ulcer disease, gastrointestinal bleeding or perforation
  6. Concomitant use of aspirin, other NSAIDS, anticoagulant or novel anticoagulant agent, pentoxifylline and probenecid
  7. Known bleeding disorders such as haemophilia, thrombocytopenia
  8. Heart failure
  9. Per-operative period of coronary artery bypass graft (CABG) surgery
  10. Concurrent asthmatic attack

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
The change in pain intensity over 60 mins in terms of 100-mm VAS | Measure at baseline and at 5, 15, 30 and 60 minutes after drug administration
  Patients are instructed to complete a questionnaire with visual analogue scale (VAS), a 100-mm horizontal straight line whereas"0" at the left end indicates "no pain at all" and "10" at the right end indicates "the worst possible pain I can imagine".

SECONDARY OUTCOMES:
Blood pressure | Measure at baseline and at 5, 15, 30 and 60 minutes after drug administration
  Blood pressure in mmHg
Pulse Rate | Measure at baseline and at 5, 15, 30 and 60 minutes after drug administration
  Pulse Rate in beat per minute
Oxygen saturation | Measure at baseline and at 5, 15, 30 and 60 minutes after drug administration
  Oxygen saturation in %
Level of sedation | Measure at baseline and at 5, 15, 30 and 60 minutes after drug administration
  Ramsay Sedation Scale 1-6. 1 indicates patient is anxious and agitated or restless, or both; 2 indicates patient is co-operative, oriented, and tranquil; 3 indicates patient responds to commands only; 4 indicates patient exhibits brisk response to light glabellar tap or loud auditory stimulus; 5 indicates patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus; 6 indicates patient exhibits no response.
Drug-related adverse events | After drug administration until the end of the observation period (1 hour)
  Patients are advised to report any discomfort any time during the study period. The investigator would judge whether the complaint is drug-related and give corresponding treatment. If the patients have no active complaint, they would be asked on a checklist for possible related adverse events before discharge. The nature and severity of adverse events would be documented. To exclude any late effects, discharged patients are encouraged to return to the department if they experience any adverse events.
Use of rescue medication | After drug administration until the end of the observation period (1 hour)
  Analgesics given after study drug administration in either group are considered as rescue medication. It will be given any if the patient requests or pain improvement is insufficient based on judgement of the attending physician. The name of rescue medication, dosage, time and route of administration will be documented.
Level of patient's satisfaction | After drug administration until the end of the observation period (1 hour)
  Patients are instructed to rate the overall efficacy and acceptance of the drug by five-point Likert scale on a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Ying Wong, MB ChB, Principal Investigator — Hospital Authority, Hong Kong
Locations (1):
- Hospital Authority, Hong Kong, Hong Kong